CLINICAL TRIAL: NCT02674074
Title: Evaluation of Corneal Temperature by Infrared Thermography in Glaucoma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EKNZ 120/11
Record Dates: First submitted 2016-01-27; First posted 2016-02-04 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- measurement of corneal temperature by infrared thermography (Experimental)
  Interventions: Device: infrared thermography

INTERVENTIONS:
Device: infrared thermography — measurement of corneal temperature by infrared thermography before and after cold provocation

SUMMARY:
Measurement of corneal temperature gives indirect information about the ocular blood flow. For this reason corneal temperature can be used as a surrogate to quantify ocular blood flow. It can be measured by means of infrared thermography. This test, however, is not used in an everyday clinical routine so far. In this study is investigated if ocular blood flow disturbances in glaucoma patients can be diagnosed by means of infrared thermography.

Corneal temperature are measured in normal tension glaucoma patients and healthy controls before and after cold provocation test. In the group of patients and the group of controls, subjects with and without a primary vascular dysregulation (PVD) are included. This will allow to analyze and compare the influence of cold provocation on corneal temperature (and indirectly ocular blood flow) in these study Groups.

ELIGIBILITY:
Inclusion Criteria for Patients:

* Glaucoma
* Age 18-65

Exclusion Criteria for patients:

* No Glaucoma
* Alcohol consumption
* Smoking

Inclusion Criteria for Control:

* No Glaucoma
* Age 18-65

Exclusion Criteria for control:

* Alcohol consumption
* Smoking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Corneal temperature measurement by infrared thermography | 2 measurements with interval of 5 minutes starting at baseline
  measurement of change in corneal temperature starting with first measurement at Baseline and second measurement after 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Josef Flammer, Prof. MD, Study Chair — University Hospital, Basel, Switzerland
Locations (1):
- Department of Ophthalmology, University Hospital Basel, Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No